CLINICAL TRIAL: NCT04146272
Title: A Comparative, Controlled Clinical Investigation of a New Acoustic Feedback Cancellation Strategy in Comparison With the Currently Marketed System
Brief Title: A Comparison of a New Acoustic Feedback Canceller in Hearing Aids With the Current System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bernafon AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BF004-1901
Record Dates: First submitted 2019-10-10; First posted 2019-10-31 (Actual); Results first posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-08

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: The participants will wear hearing aids with the current feedback system and the new feedback system each for 10 +/- 5 days. Some will wear the current hearing aids first and some will wear the new Hearing aids first.
Who Masked: Participant
Masking Description: The participants are masked during the lab testing. They will not know which device they are testing because the Investigator will place it on their ear without letting them see it.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Moderate Hearing loss current Mermaid first, then new (Active Comparator): Participants were randomized to wear the current Mermaid hearing aid that uses the current feedback cancellation first for 10 days. Then they wore the new Mermaid Hearing aid for another 10 days.
  Interventions: Device: Hearing Aid Mermaid Current; Device: Hearing Aid Mermaid New
- Moderate Hearing loss new Mermaid first, then current (Active Comparator): Participants were randomized to wear the new Mermaid hearing aid that uses the new feedback cancellation first for 10 days. Then they wore the current Mermaid Hearing aid for another 10 days.
  Interventions: Device: Hearing Aid Mermaid Current; Device: Hearing Aid Mermaid New
- Severe hearing loss current Power first, then new (Active Comparator): Participants were randomized to wear the current power hearing aid that uses the current feedback cancellation first for 10 days. Then they wore the new power Hearing aid for another 10 days.
  Interventions: Device: Power Hearing Aid Current; Device: Power Hearing Aid New
- Severe hearing loss new Power first, then current (Active Comparator): Participants were randomized to wear the new power hearing aid that uses the new feedback cancellation first for 10 days. Then they wore the current power Hearing aid for another 10 days.
  Interventions: Device: Power Hearing Aid Current; Device: Power Hearing Aid New

INTERVENTIONS:
Device: Hearing Aid Mermaid Current — The current hearing aid used to treat hearing loss.
  Arms: Moderate Hearing loss current Mermaid first, then new; Moderate Hearing loss new Mermaid first, then current
Device: Hearing Aid Mermaid New — The new hearing aid used to treat hearing loss with an upgraded feedback cancellation system.
  Arms: Moderate Hearing loss current Mermaid first, then new; Moderate Hearing loss new Mermaid first, then current
Device: Power Hearing Aid Current — The current power hearing aid used to treat strong hearing loss.
  Arms: Severe hearing loss current Power first, then new; Severe hearing loss new Power first, then current
Device: Power Hearing Aid New — The new power hearing aid used to treat strong hearing loss with an upgraded feedback cancellation system.
  Arms: Severe hearing loss current Power first, then new; Severe hearing loss new Power first, then current

SUMMARY:
The Purpose of the study is to show that the performance of the new feedback cancellation system is better than the feedback system used in the currently marketed hearing aids. Speech understanding should not be negatively affected by the new system, ad there should be no consequential artifacts or unwanted noises caused by the new system.

DETAILED DESCRIPTION:
The amplification of sounds with a hearing aid is the most common treatment for hearing loss. Benefits of amplification and accessories used with it outweigh any risks in mild to profound hearing-impaired subjects. Hearing aids provide a benefit for people with only a mild sensorineural hearing loss. However, often people are counselled to wait to purchase hearing aids until their hearing loss becomes more significant. The benefits are obtainable for both unilateral and bilateral fittings and are both short term and durable on long term.

Acoustic feedback is a critical problem to all hearing aids. The acoustic coupling between the hearing aid receiver and the microphone occurs when an endless loop is formed so that the microphone is re-amplifying sound from its own receiver. The higher the amplification of the system, the more unstable it becomes and the more likely an acoustic feedback will occur. When this happens the hearing aid user and those around them hear a loud whistling noise. A common method used to combat this problem is feedback cancellation, more specifically adaptive feedback cancellation. The goal of feedback cancellation is to quickly identify feedback path changes and make adjustments to preserve the stability of the system while maintaining a high sound quality and still providing a high stable gain compared to the gain achieved without an active feedback reduction.

For this study, the Sponsor will carry out testing with participants who have hearing loss to validate the performance of the new feedback cancelling algorithm. Studies have investigated the advantages and disadvantages of different feedback cancellation techniques. However, it is accepted by professionals that having a feedback system is better than not using feedback cancellation. The Sponsor has used an adaptive feedback cancellation algorithm since 2010. For the current study the new adaptive algorithm will be compared to the current algorithm implemented in the hearing aids that are certified by the European Conformity and sold on the market. The aim is to determine if less feedback is experienced using the new system in comparison to the old system.

ELIGIBILITY:
Inclusion Criteria:

* All classifications of hearing loss (sensorineural, conductive, mixed)
* Conductive and mixed hearing loss must be approved for amplification by a physician
* All shapes of hearing loss (flat, sloping, reverse slope, notch)
* Severity ranging from mild to profound
* German speaking
* Ability and willingness to sign the consent form

Exclusion Criteria:

* Contraindications for amplification
* Active ear disease
* New hearing aid users
* Inability to follow the procedures
* Reduced mobility that makes then unable to attend study Appointments
* Uncooperative so that it's not possible to get a valid audiogram
* A strongly reduced dexterity
* Central hearing disorder
* Sponsor employees
* Family members of Sponsor employees

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Babara Simon, AuD, Principal Investigator — Sponsor/Bernafon
Locations (1):
- Bernafon, Bern, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 33 patients were screened for eligibility from the list of contacts at the Bernafon Hearing clinic.
Pre-assignment Details: 33 participants were randomized. 22 met the inclusion criteria for moderate Hearing loss and 11 for severe Hearing loss.
Groups:
- Moderate Hearing Loss Current Mermaid, Then New: Participants first used the current Mermaid hearing aid with the current feedback cancellation system for 10 days. Then they used the new Mermaid Hearing aid with the new feedback system for 10 days.
- Moderate Hearing Loss New Mermaid, Then Current: Participants first used the new Mermaid hearing aid with the new feedback cancellation system for 10 days. Then they used the current Mermaid Hearing aid with the current feedback system for 10 days.
- Severe Hearing Loss Current Power, Then New: Participants first used the current power hearing aid with the current feedback cancellation system for 10 days. Then they used the new power Hearing aid with the new feedback system for 10 days.
- Severe Hearing Loss New Power First/Current Second: The new power hearing aid that is not yet sold and uses the new feedback cancellation system will be worn first by this group. The current power hearing aid that is sold and uses the current feedback cancellation system will be used as a comparator and worn second.
Period: First Intervention
Arm/Group | Moderate Hearing Loss Current Mermaid, Then New | Moderate Hearing Loss New Mermaid, Then Current | Severe Hearing Loss Current Power, Then New | Severe Hearing Loss New Power First/Current Second
Started | 11 | 11 | 6 | 5
Completed | 11 | 11 | 6 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Second Intervention
Arm/Group | Moderate Hearing Loss Current Mermaid, Then New | Moderate Hearing Loss New Mermaid, Then Current | Severe Hearing Loss Current Power, Then New | Severe Hearing Loss New Power First/Current Second
Started | 11 | 11 | 6 | 5
Completed | 11 | 11 | 6 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Mermaid group included Hearing impaired with a mild to severe Hearing loss and a mean age of 67. The Power group included Hearing impaired with a moderate to profound Hearing loss and a mean age of 67.
Groups:
- Current Mermaid First, Then New: Participants were randomized to wear the current hearing aid that uses the current feedback cancellation first for 10 days. Then they wore the new Hearing aid for another 10 days.
- New Mermaid First, Then Current: Participants were randomized to wear the new Hearing aid that uses the new feedback cancellation first for 10 days. Then they wore the current Hearing aid for another 10 days.
- Current Power First, Then New: Participants were randomized to wear the current power hearing aid that uses the current feedback cancellation first for 10 days. Then they wore the new power Hearing aid for another 10 days.
- New Power First, Then Current: Participants were randomized to wear the new power hearing aid that uses the new feedback cancellation first for 10 days. Then they wore the current power Hearing aid for another 10 days.
- Total: Total of all reporting groups
Arm/Group | Current Mermaid First, Then New | New Mermaid First, Then Current | Current Power First, Then New | New Power First, Then Current | Total
Number analyzed (Participants) | 11 | 11 | 6 | 5 | 33
Age, Continuous [Mean (Full Range); unit: years] | 67 [38 to 74] | 67 [45 to 80] | 67 [49 to 79] | 67 [57 to 86] | 67 [38 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 1 | 8
  Male | 9 | 8 | 4 | 4 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Switzerland | 11 | 11 | 6 | 5 | 33
Hearing Threshold [Mean (Standard Deviation); unit: decibels] — The threshold is the lowest/softest tone measured in decibels (dB) that a Person can hear during the testing and it measured at various frequencies from 250 to 8000 Hertz (Hz). The louder that the tone Needs to be in order to hear it, the more Hearing loss that a Person has.
  decibels | 47 (11.7) | 50 (13.1) | 69 (10.2) | 71 (10.6) | 59 (11)

OUTCOME MEASURES:

1. Primary Outcome: Change in Live Feedback Test Scores From Day 10 to Day 20
Description: In the lab, subjects will have the hearing aid placed in their ear. They will rate on a visual analogue scale whether feedback occurs and if so, how much annoyance it causes. The scale has a minimum of 0 and a maximum of 10. A lower score is a better answer. It will be tested in two conditions, aided with the current Hearing aid, and aided with the new Hearing aid at 10 and 20 days. The difference between the scores from day 10 and day 20 was calculated by subtracting day 20 ("new hearing aid") from day 10 ("current hearing aid") after both sessions of testing were completed and reported as the mean difference for the group. Regardless of the arm assignment, participants wore the same hearing aids for the lab test on days 10 and 20.
Time Frame: 10 days, 20 days
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Moderate Hearing Loss Current Mermaid First/New Second: The current Mermaid hearing aid that is sold and uses the current feedback cancellation system will be used as a comparator and worn first for this group. The new Hearing aid with the new feedback system will be used second.
- Moderate Hearing Loss New Mermaid First/Current Second: The new Mermaid Hearing aid with the new feedback system will be worn first for this group.The current hearing aid that is sold and uses the current feedback cancellation system will be used as a comparator and worn second.
- Severe Hearing Loss Current Power First/New Second: The current power hearing aid that is sold and uses the current feedback cancellation system will be used as a comparator and worn first by this group. The new power hearing aid that is not yet sold and uses the new feedback cancellation system will be worn second.
Arm/Group | Moderate Hearing Loss Current Mermaid First/New Second | Moderate Hearing Loss New Mermaid First/Current Second | Severe Hearing Loss Current Power First/New Second | Severe Hearing Loss New Power First/Current Second
Number analyzed (Participants) | 11 | 11 | 6 | 5
units on a scale | 1.7 (2.0) | 1.7 (2.0) | 0.1 (1.1) | 0.1 (1.1)

2. Secondary Outcome: Word Recognition - Aided
Description: Subjects will indicate on a touch screen which word that they heard through the loud speaker. The touch screen will give 5 possible answer choices that includes the correct choice and 4 other words that rhyme with the actual word. The test is run in the aided condition with the current Hearing aid and with the new Hearing aid. The test is scored by the percentage of words that they answer correctly. 0 percent is the lowest score possible and 100 percent is the highest. A higher percentage indicates a better score.
Time Frame: 20 days
Measure: Mean (Standard Deviation); unit: percentage of words correct
Arm/Group | Moderate Hearing Loss Current Mermaid First, Then New | Moderate Hearing Loss New Mermaid First, Then Current | Severe Hearing Loss Current Power First, Then New | Severe Hearing Loss New Power First, Then Current
Number analyzed (Participants) | 11 | 11 | 6 | 5
percentage of words correct
  Current hearing | 0.92 (0.34) | 0.92 (0.34) | 0.77 (0.49) | 0.77 (0.49)
  New hearing aid | 0.91 (0.35) | 0.91 (0.35) | 0.78 (0.48) | 0.78 (0.48)

3. Secondary Outcome: Sound Quality Rating
Description: The subjects will complete a questionnaire that asks them to rate the quality of different aspects of the hearing aid including sound quality, own voice quality, and the sound quality when in a noisy environment. The scale is from 1 to 5 with 1 being the minimum and 5 being the maximum. A higher score indicates better quality.
  The questionnaire will be answered for two conditions, aided with the current Hearing aid and aided with the new Hearing aid. The difference between the scores for each condition will be calculated and reported as the mean difference across both arms (moderate hearing loss and severe hearing loss). The difference is not calculated over time points but at the end of the field trial and the assignment order of the hearing aid (new first or current first) does not bear an impact.
Time Frame: 20 days
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Severe Hearing Loss New Power First/Current Second: Participants were randomized to wear the new power hearing aid that uses the new feedback cancellation first for 10 days. Then they wore the current power Hearing aid for another 10 days.
Arm/Group | Moderate Hearing Loss Current Mermaid First, Then New | Moderate Hearing Loss New Mermaid First, Then Current | Severe Hearing Loss Current Power First, Then New | Severe Hearing Loss New Power First/Current Second
Number analyzed (Participants) | 11 | 11 | 6 | 5
units on a scale | 1.6 [1.0 to 2.1] | 1.6 [1.0 to 2.1] | 1.5 [0.1 to 2.9] | 1.5 [0.1 to 2.9]

4. Other Pre Specified Outcome: Number of Participants Reporting an Adverse Event
Description: The safety of the hearing aids will be rated by the number of adverse events reported by subjects. The minimum score is Zero and the maximum is not defined but is likely not more than 20. A lower number of adverse Events indicates a better outcome. The Outcome will be reported as the sum of Adverse Events reported across time frames.
Time Frame: 0, 10, and 20 days
Measure: Count of Participants; unit: Participants
Groups:
- Moderate Hearing Loss Current Mermaid Hearing Aid: Participants with a moderate hearing loss that reported an AE while wearing the Mermaid hearing aid that uses the current feedback cancellation regardless of randomization order.
- Moderate Hearing Loss New Mermaid Hear Aid: Participants with a moderate hearing loss that reported an AE while wearing the Mermaid hearing aid that uses the new feedback cancellation regardless of randomization order.
- Severe Hearing Loss Current Power Hear Aid: Participants with a severe hearing loss that reported an AE while wearing the current Power hearing aid regardless of randomization order.
- Severe Hearing Loss New Power Hearing Aid: Participants with a severe hearing loss that reported an AE while wearing the new Power hearing aid regardless of randomization order.
Arm/Group | Moderate Hearing Loss Current Mermaid Hearing Aid | Moderate Hearing Loss New Mermaid Hear Aid | Severe Hearing Loss Current Power Hear Aid | Severe Hearing Loss New Power Hearing Aid
Number analyzed (Participants) | 5 | 3 | 1 | 3
Participants | 5 | 3 | 1 | 3

5. Secondary Outcome: Word Recognition - Unaided
Description: This measurement is made without any hearing aids. Subjects will indicate on a touch screen which word that they heard through the loud speaker. The touch screen will give 5 possible answer choices that includes the correct choice and 4 other words that rhyme with the actual word. The test is run in the unaided condition. The test is scored by the percentage of words that they answer correctly. 0 percent is the lowest score possible and 100 percent is the highest. A higher percentage indicates a better score. The scores are not dependent on the assignment order of the hearing aids (new or current first) as the measurement is made without hearing aids and a score calculated for each group (moderate or severe hearing loss) and not for each arm.-
Time Frame: 10 days
Measure: Mean (Standard Deviation); unit: percentage of words correct
Arm/Group | Moderate Hearing Loss Current Mermaid First, Then New | Moderate Hearing Loss New Mermaid First, Then Current | Severe Hearing Loss Current Power First, Then New | Severe Hearing Loss New Power First, Then Current
Number analyzed (Participants) | 11 | 11 | 6 | 5
percentage of words correct | 0.79 (0.48) | 0.79 (0.48) | 0.40 (0.58) | 0.40 (0.58)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: The Definition is the same. The participants are asked at every Appointment about any Events that may have occurred during the time since the last Appointment.
Groups:
- Moderate Hearing Loss Current Mermaid Hearing Aid: The number of participants with a moderate hearing loss to report an AE while wearing the Mermaid hearing aid with the current feedback system regardless of the randomization order.
- Moderate Hearing Loss New Mermaid Hearing Aid: The number of participants with a moderate hearing loss to report an AE while wearing the Mermaid hearing aid with the new feedback system regardless of the randomization order.
- Severe Hearing Loss Current Power Hearing Aid: The number of participants with a severe hearing loss to report an AE while wearing the current Power hearing aid regardless of the randomization order.
- Severe Hearing Loss New Power Hearing Aid: The number of participants with a severe hearing loss to report an AE while wearing the new Power hearing aid regardless of the randomization order.
Arm/Group | Moderate Hearing Loss Current Mermaid Hearing Aid | Moderate Hearing Loss New Mermaid Hearing Aid | Severe Hearing Loss Current Power Hearing Aid | Severe Hearing Loss New Power Hearing Aid
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 5/22 | 3/22 | 1/11 | 3/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moderate Hearing Loss Current Mermaid Hearing Aid (N=22) | Moderate Hearing Loss New Mermaid Hearing Aid (N=22) | Severe Hearing Loss Current Power Hearing Aid (N=11) | Severe Hearing Loss New Power Hearing Aid (N=11)
Cold (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) — Common cold that did not Need Treatment.
Bodily harm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Subjects suffered an accident and injured a part of the body but required no Treatment.
Skin irritation (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) — Subjects had a skin irritation that required no treatment
Pain (Product Issues) | 1 (1) | 1 (1) | 0 (0) | 2 (2) — Subjects reported pain that required no treatment

LIMITATIONS AND CAVEATS:
No limitations or caveats

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-09-13): https://cdn.clinicaltrials.gov/large-docs/72/NCT04146272/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/72/NCT04146272/SAP_001.pdf